CLINICAL TRIAL: NCT05721209
Title: Virtual Reality Treadmill Training in Individuals With Traumatic Brain Injur : A Pilot Study
Brief Title: Virtual Reality Treadmill Training in Individuals With Traumatic Brain Injury
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment for this study is temporarily paused due to study staff turnover.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-01576
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VRTT With Feedback - Adults (Experimental): Adults aged 18-65 with TBI. At Week 1 after baseline, participants will begin study intervention on the C-Mill with augmented/virtual reality (AR/VR) guidance. Starting at Week 2, the study intervention on C-Mill will be repeated 3 sessions/week for 8 weeks.
  Each one hour session will include about 15 minutes of standing balance training, about 5 minutes of stepping balance training and about 30 minutes of walking training on the C-Mill with AR/VR feedback.
  Interventions: Device: C-Mill with AR/VR Guidance; Device: Zeno 3-Layer Walkway; Device: Hunova
- VRTT With Feedback - Older Adults (Experimental): Adults aged 65 and older with TBI. At Week 1 after baseline, participants will begin study intervention on the C-Mill with augmented/virtual reality (AR/VR) guidance. Starting at Week 2, the study intervention on C-Mill will be repeated 3 sessions/week for 8 weeks.
  Each one hour session will include about 15 minutes of standing balance training, about 5 minutes of stepping balance training and about 30 minutes of walking training on the C-Mill with AR/VR feedback.
  Interventions: Device: C-Mill with AR/VR Guidance; Device: Zeno 3-Layer Walkway; Device: Hunova
- VRTT Without Feedback - Adults (Active Comparator): Adults aged 18-65 with TBI. At Week 1 after baseline, participants will begin study intervention on the C-Mill without augmented/virtual reality (AR/VR) guidance. Starting at Week 2, the study intervention on C-Mill will be repeated 3 sessions/week for 8 weeks.
  Each one hour session will include about 15 minutes of standing balance training, about 5 minutes of stepping balance training and about 30 minutes of walking training on the C-Mill without AR/VR feedback.
  Interventions: Device: C-Mill without AR/VR Guidance; Device: Zeno 3-Layer Walkway; Device: Hunova
- VRTT Without Feedback - Older Adults (Active Comparator): Adults aged 65 and older with TBI. At Week 1 after baseline, participants will begin study intervention on the C-Mill without augmented/virtual reality (AR/VR) guidance. Starting at Week 2, the study intervention on C-Mill will be repeated 3 sessions/week for 8 weeks.
  Each one hour session will include about 15 minutes of standing balance training, about 5 minutes of stepping balance training and about 30 minutes of walking training on the C-Mill without AR/VR feedback.
  Interventions: Device: C-Mill without AR/VR Guidance; Device: Zeno 3-Layer Walkway; Device: Hunova

INTERVENTIONS:
Device: C-Mill with AR/VR Guidance — Treadmill training system that is a combination of an instrumented treadmill, front display, and a floor projector, allowing functional gait and balance training. The AR/VR feedback will include computer generated obstacles and objects projected as images on the treadmill. Participants will be asked to use these projections as stepping cues and step on some images of objects while avoiding stepping on the images of obstacles.
  Arms: VRTT With Feedback - Adults; VRTT With Feedback - Older Adults
Device: C-Mill without AR/VR Guidance — Treadmill training system that is a combination of an instrumented treadmill, front display, and a floor projector, allowing functional gait and balance training.
  Arms: VRTT Without Feedback - Adults; VRTT Without Feedback - Older Adults
Device: Zeno 3-Layer Walkway — Used to conduct mobility assessments to assess temporal and spatial gait parameters during the 6-minute walk test.
Device: Hunova — Used to conduct fall-risk assessment.

SUMMARY:
This pilot study aims to determine the feasibility of a virtual reality treadmill training intervention in individuals with Traumatic Brain Injury (TBI). Participants will be stratified based on age into adults' group or older adults' group and then randomized into the virtual reality treadmill training (intervention) group with feedback or the treadmill training (control) group. This pilot study will also provide preliminary evidence on the impact of the virtual reality treadmill training on mobility, balance, fear of falls, fall risk, attention and physical activity in the community in individuals with TBI. The data collected in this pilot study will also help to estimate sample size for subsequent large clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 90 years old
2. diagnosed with a non-penetrating TBI
3. at least 12 months post most recent injury
4. self-reported balance deficits and fear of falls or at least 2 falls in the last one year
5. Able to understand and speak English language to respond, understand and comply with study procedures throughout the 10-week study period and fill out the study questionnaires in English
6. Able to walk with minimal assistance or less (with bracing and assistive devices as needed)

Exclusion Criteria:

1. history of severe cardiac disease
2. neuromuscular or neurological pathologies other than TBI that limit study participation
3. uncontrolled seizure disorder
4. weight greater than 135 kg or less than 25 kg
5. height greater than 6' 2''
6. severe cognitive, visual or hearing impairment where the patient is not able to follow the study instructions
7. open skin lesion or bandage in the area of C-Mill harness contact

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2026-12-23 (Estimated); Study Completion 2026-12-23 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Up to Week 10
  Recruitment rate is defined as the number of patients recruited on average for one month in one site.
Enrollment Rate | Up to Week 10
  Enrollment Rate defined as the percentage of recruited participants who enrolled in the study.
Retention Rate | Up to Week 10
  Retention rate defined as the percentage of enrolled participants who completed the study.
Percentage of Participants who Adhere to 100% of Study Procedures | Up to Week 10

SECONDARY OUTCOMES:
Change from Baseline in Falls Self-Efficacy Scale (FES-I) Score by Final Intervention Visit | Baseline, Week 7
  FES-I is a 16-item self-assessment of fear of falls in different situations. Each item is ranked on a 4-point Likert scale ranging from 1 (Not at all concerned) to 4 (Very concerned). The total score is the sum of responses and ranges from 16 to 64; lower scores indicate lower fear of falls. A decrease in scores indicates fear of falls decreased over the observational period.

CONTACTS AND LOCATIONS:
Overall Officials: Akhila Veerubhotla, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Shared data will be aggregated and deidentified. No IPD will be shared with other researchers.